CLINICAL TRIAL: NCT03116984
Title: A Prospective, Randomized, Multicenter Study of Comparison of TACE Combination With and Without EBRT for HCC Which is Unresectable But Confined to the Liver
Brief Title: A Study of Comparison of TACE Combination With and Without EBRT for Advanced HCC
Acronym: TACE-EBRT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Changhai Hospital (Other); Shanghai 10th People's Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Fujian Cancer Hospital (Other Government); First Affiliated Hospital of Fujian Medical University (Other); Zhongshan Hospital Xiamen University (Other); West China Hospital (Other); Peking University Cancer Hospital & Institute (Other); Xinqiao Hospital of Chongqing (Other); 309th Hospital of Chinese People's Liberation Army (Other); Heilongjiang Provincial Agricultural Reclamation General Hospital (Unknown); Longyan First Hospital, Affiliated to Fujian Medical University (Unknown); Peking University First Hospital (Other); The Third Affiliated Hospital of Qiqihar Medical Universitiy (Unknown); Anhui Provincial Hospital (Other Government); First Affiliated Hospital of Xinjiang Medical University (Other); Qingdao University (Other); The 4th people's hospital of Wuxi City, Affiliated to Jiangnan University (Unknown); Subei People's Hospital of Jiangsu Province,Yangzhou University (Unknown); Affiliated Zhongshan Hospital of Dalian University (Other); Jilin University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Fudan University (Other); Shanghai East Hospital,Tongji University School of Medicine (Unknown); Chinese PLA General Hospital (Other); The 4th People's Hospital of Linfen City (Unknown); Nanfang Hospital, Southern Medical University (Other); Yunnan Cancer Hospital (Other); Shandong Cancer Hospital and Institute (Other); Sichuan Cancer Hospital and Research Institute (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); Fujian Medical University Union Hospital (Other); The People's Hospital of Hunan Province (Unknown)
Responsible Party: Principal Investigator, Zeng Zhaochong, Director, Head of Department of Radiation Oncology, Principal Investigator, Clinical Professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZS-TACE-EBRT-2017; 2016ZSLC20 (Other Grant/Funding Number: Zhongshan Hospital, Fudan University)
Record Dates: First submitted 2017-03-01; First posted 2017-04-17 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; external- beam radiotherapy (EBRT); transarterial chemoembolization (TACE)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcatheter arterial chemoembolization (Active Comparator): TACE group: The frequency of treatment is determined based on the disease condition for patients who are randomly assigned to group of TACE treatment.TACE is performed via an injection into the hepatic artery of agents by puncturing the common femoral artery, and micro-embolization superselective catheterization is preferred.Adriamycin(30 to 60mg) is considered as basic chemotherapy drugs in the process of transcatheter endovascular perfusion.The dose of ultra fluid lipiodol was determined by diameter and blood supply type of HCC,generally 5-20ml, and no more than 30ml once.The boundary is considered whether there are large amounts of lipiodol to deposit in the tumor and tiny branches shadow of portal veins in paracarcinoma under fluoroscopic guidance. Embolizing agents(gelatin sponge particles 350um-560um) are added after lipiodol emulsion embolization.It has a possibility of observeation alone if tumor achieves a complete response after two times TACE.
  Interventions: Procedure: Transcatheter arterial chemoembolization
- External-beam radiotherapy (Experimental): EBRT group: Patients who were randomized to the external- beam radiotherapy (EBRT) 3-5 weeks after the completion 2 times TACE.Radiotherapy equipment is based on the conditions of the cooperative units. 3-DCRT, IMRT or IGRT will be opted based on hospital. IGRT can also be used via helical tomotherapy, Rapid Arc or VMAT. The target volume should include the visible tumor.
  Interventions: Radiation: External- beam radiotherapy

INTERVENTIONS:
Procedure: Transcatheter arterial chemoembolization — Transcatheter arterial chemoembolization (TACE) is performed via an injection into the hepatic artery of agents by puncturing the common femoral artery.Adriamycin(30 to 60 mg) is considered as basic chemotherapy drugs in the process of transcatheter endovascular perfusion. The dose of lipiodol was determined by diameter and blood supply type of HCC, generally 5-20ml, and no more than 30ml once.
  Other Names: TACE
  Arms: Transcatheter arterial chemoembolization
Radiation: External- beam radiotherapy — We have reported a series of retrospective clinical trials in which transarterial chemoembolization (TACE) combined with external- beam radiotherapy (EBRT) was a better treatment method than TACE alone for unresectable HCC in the same period and organization, no matter in aspects of the regression rate of carcinoma or survival.Patients who were randomized to the EBRT 3-5 weeks after the completion 2 times TACE.
  Other Names: EBRT
  Arms: External-beam radiotherapy

SUMMARY:
This clinical trial is a prospective, randomized, controlled and multicenter study.And the trial is going to better control intrahepatic tumors for hepatocellular carcinoma(HCC) patients who meet the inclusion criterion.The patients were divided into two groups, the group A by TACE and the other group B by external- beam radiotherapy(EBRT) after 2 times TACE. Then the therapeutic effects and toxicities of TACE and EBRT are evaluated during the follow-up period. The study design plans to enroll 300 patients, and each group includes 150 cases.

DETAILED DESCRIPTION:
Enrolled HCC patients met the inclusion criterion, in the late or advanced stage,tumor confined in intrahepatic( meet the tolerance-dose for the liver), without cancer embolus in main branch of portal vein, without extrahepatic metastasis and the number of tumor was≤3. Eligible participants will be randomly assigned to the group A by TACE and the other group B by EBRT after 2 times TACE.

TACE group: The frequency of treatment is determined based on the disease condition for patients who are randomly assigned to group of TACE.TACE is performed via an injection into the hepatic artery of agents by puncturing the common femoral artery, and micro-embolization superselective catheterization is preferred.Adriamycin(30 to 60mg) is considered as basic chemotherapy drugs in the process of transcatheter endovascular perfusion.The dose of fluid lipiodol was determined by diameter and blood supply type of HCC,generally 5-20ml, and no more than 30ml once.The boundary is considered whether there are large amounts of lipiodol to deposit in the tumor and tiny branches shadow of portal veins in paracarcinoma under fluoroscopic guidance. Embolizing agents(gelatin sponge particles 350um-560um) are added after lipiodol emulsion embolization.It has a possibility of observeation alone if tumor achieves a complete response after two times TACE.

EBRT group: Patients who were randomized to the radiotherapy group start radiotherapy 3-5 weeks after the completion 2 times TACE and began to undergo radiation. Radiotherapy equipment is based on the conditions of the cooperative units. 3-dimensional conformal radiation therapy(3-DCRT), intensity-modulated radiation therapy(IMRT) or Image-Guided Radiotherapy(IGRT) will be opted based on hospital. IGRT can also be used via helical tomotherapy, Rapid Arc or Volumetric Modulated Arc Therapy(VMAT). The target volume should include the visible tumor.

ELIGIBILITY:
1. Inclusion Criteria 1）initially diagnosed HCC (confirmed by pathology or meet clinical diagnostic criteria), 2）The patients are not candidates for curative surgery, which should be determined in consultation with two oncology surgeons of the same center, 3）Tumor was confined in intrahepatic( meet the tolerance-dose for the liver), without cancer embolus in main branch of portal vein, without extrahepatic metastasis and the number of tumor was≤3, 4）Child-Pugh A，white blood cell count >2*109/L、Hb>90g/L、PLT>50*109/L, 5）The score of Eastern Cooperative Oncology Group(ECOG): 0-2, 6）The estimated survival time > 3 months, 7）Without midsection history of radiation therapy, 8）Age: >18 years old, 9）Informed consent was signed.
2. Exclusion Criteria 1）Diffuse hepatocellular carcinoma, 2）Uncontrollable infection, 3）Concurrent other malignant tumors, 4）Simultaneously participate in other experimental drugs or clinical trials, 5）Serious of heart, lung and kidney diseases, 6）During pregnancy and lactation, 7) The ones with severe neurologic morbidity couldn't clearly tell therapeutic response.
3. Halfway exit criteria 1）Do not treat according to the research or seriously violate the fundamental principles after enrolled, 2）Cannot tolerate radiation therapy, including the ones that cann't complete the radiation treatment( the dose <40 Gy,biological effective dose <48 Gy), or interrupt more than 2 weeks during radiotherapy, 3）Unwilling to continue this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival(OS) | The outcome measures are assessed up to three years.
  The therapeutic effects are mainly evaluated by the 3-year overall survival(OS).

CONTACTS AND LOCATIONS:
Overall Officials: Zhongshan Hospital, Study Director — Fudan University, Shanghai, China
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No